CLINICAL TRIAL: NCT02122367
Title: Validation of Stroke Volume Variation and Pleth Variability Index as Predictors of Fluid Responsiveness in Patients Undergoing Robot Assisted Thyroidectomy
Brief Title: Study of Stroke Volume Variation and Pleth Variability Index as Predictors of Fluid Responsiveness
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, So Young Yang, So young Yang MD,PhD, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Chung-Ang UH
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Thyroidectomy; Fluid Responsiveness
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives

ARMS (1):
- stroke volume variation, pleth variability index (Experimental): stroke volume variation: recorded using the FloTrac/Vigileo system (Edwards Lifesciences)
  pleth variability index: recorded using the Masimo Radical-7 monitor (Masimo Corporation, Irvine, CA, USA)
  Interventions: Other: HES 130/0.4 (VolulyteⓇ, Fresenius Kabi, Canada)

INTERVENTIONS:
Other: HES 130/0.4 (VolulyteⓇ, Fresenius Kabi, Canada) — HES 130/0.4 (VolulyteⓇ, Fresenius Kabi, Canada) 6ml/kg of ideal body weight loading

SUMMARY:
Appropriate indices to guide fluid therapy are essential for effective hemodynamic management during the perioperative period. Values derived from respiratory changes in arterial pressure waveform or plethysmographic waveform such as stroke volume variation and pleth variability index have been demonstrated to be able to predict fluid responsiveness in surgical or critically ill patients. Their ability to predict fluid responsiveness can be affected by factors that influence the arterial tone or the compliance of the respiratory system by position change. The aim of this prospective trial is to investigate the ability of stroke volume variation and pleth variability index to predict fluid responsiveness in the reverse trendelenberg position.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20
2. elective robot assisted thyroidectomy

Exclusion Criteria:

1. arrhythmia
2. BMI>30
3. valvular heart disease
4. pul hypertension
5. peripheral artery occlusive disease
6. lung disease
7. right heart failure

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
stroke volume variation | 5 minutes after volume replacement
pleth variability index | 5 minutes after volume replacement

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Seoul, Seoul, South Korea